CLINICAL TRIAL: NCT03037385
Title: A Phase 1/2 Study of the Highly-selective RET Inhibitor, BLU-667, in Patients With Thyroid Cancer, Non-Small Cell Lung Cancer (NSCLC) and Other Advanced Solid Tumors
Brief Title: Phase 1/2 Study of the Highly-selective RET Inhibitor, Pralsetinib (BLU-667), in Participants With Thyroid Cancer, Non-Small Cell Lung Cancer, and Other Advanced Solid Tumors
Acronym: ARROW
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO42863; 2016-004390-41 (EudraCT Number); BLU-667-1101 (Registry Identifier: CT.Gov)
Expanded Access: NCT04204928 (Approved for marketing)
Record Dates: First submitted 2017-01-20; First posted 2017-01-31 (Estimated); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: RET-altered Non Small Cell Lung Cancer; Medullary Thyroid Cancer; RET-altered Papillary Thyroid Cancer; RET-altered Colon Cancer; RET-altered Solid Tumors; Lung Neoplasm; Carcinoma, Non-Small-Cell Lung; Thyroid Diseases; Thyroid Neoplasm; Thyroid Cancer, Papillary; Carcinoma, Neuroendocrine; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Disease; Carcinoma, Bronchogenic; Bronchial Neoplasms; Endocrine System Diseases; Endocrine Gland Neoplasm; Head and Neck Neoplasms; Adenocarcinoma, Papillary; Adenocarcinoma; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neuroendocrine Tumors; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms, Nerve Tissue; Colonic Neoplasms; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasm; Digestive System Disease; Gastrointestinal Disease; Colonic Diseases; Intestinal Disease
Keywords: RET Lung; RET Thyroid; RET fusion; RET alteration; RET mutation; RET positive; RET inhibitor; RET altered; RET rearrangement; RET NSCLC; RET medullary thyroid cancer; RET-rearranged NSCLC; RET-rearranged thyroid; M918T; TRIM33-RET; RET fusion lung cancer; RET fusion thyroid cancer; lung cancer mutation; BLU 667; RET tyrosine kinase; RET gene mutation; RET kinase; RET MTC; advanced lung cancer; advanced non small cell lung cancer; metastatic lung cancer; KIF5B-RET; CCDC6-RET; NCOA4-RET; advance solid tumor; V804L; V804M; thyroid cancer RET inhibitor; lung cancer RET inhibitor; RET PTC; rearranged during transfection; RET-PTC1; RET-PTC; RET-PTC3; RET-PTC4; PRKAR1A-RET; RET-PTC2; GOLGA5-RET; RET-PTC5; ERC1-RET; KTN1-RET; RET-PTC8; HOOK3-RET; PCM1-RET; TRIM24-RET; RET-PTC6; TRIM27-RET; RET-PTC7; AKAP13-RET; FKBP15-RET; SPECC1L-RET; TBL1XR1-RET; BCR-RET; FGRF1OP-RET; RFG8-RET
MeSH Terms: conditions — Carcinoma, Medullary; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Thyroid Diseases; Thyroid Neoplasms; Thyroid Cancer, Papillary; Carcinoma, Neuroendocrine; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Endocrine System Diseases; Endocrine Gland Neoplasms; Head and Neck Neoplasms; Adenocarcinoma, Papillary; Adenocarcinoma; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neuroendocrine Tumors; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms, Nerve Tissue; Colonic Neoplasms; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Multiple Endocrine Neoplasia Type 2a | interventions — pralsetinib

STUDY DESIGN:
Intervention Model Description: Phase 1 (Complete):
  * Advanced MTC, NSCLC or other solid tumor
  * 30-600mg (PO QD or BID)
  Phase 2 (400mg QD):
  * Group 1: RET fusion NSCLC previously treated with a platinum chemotherapy
  * Group 2: RET fusion NSCLC not previously treated for metastatic disease
  * Group 3: MTC previously treated with cabozantinib and/or vandetanib
  * Group 4: MTC not previously treated with cabozantinib or vandetanib
  * Group 5: Other solid tumors with a RET fusion not eligible for any of the other groups and previously treated with SOC or have no acceptable SOC for their tumor type as determined by the investigator
  * Group 6: Any solid tumor with a RET alteration (fusion or mutation) previously treated with a selective RET Inhibitor
  * Group 7: Other solid tumors with a RET mutation previously treated with SOC
  * Group 8: RET fusion NSCLC previously treated with a platinum chemotherapy (China only)
  * Group 9: MTC not previously treated with systemic therapy for advanced or metastatic disease (China only)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose Escalation (Experimental): Multiple doses of pralsetinib (BLU-667) for oral administration.
  Interventions: Drug: pralsetinib (BLU-667)
- Phase 2 Dose Expansion (Experimental): Oral dose of pralsetinib (BLU-667) as determined during Dose Escalation.
  Interventions: Drug: pralsetinib (BLU-667)

INTERVENTIONS:
Drug: pralsetinib (BLU-667) — pralsetinib (BLU-667) is a potent and selective inhibitor of the RET mutations, fusions, and predicted resistant mutants
  Other Names: BLU-667

SUMMARY:
This is a Phase 1/2, open-label, first-in-human (FIH) study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antineoplastic activity of pralsetinib (BLU-667) administered orally in participants with medullary thyroid cancer (MTC), RET-altered NSCLC and other RET-altered solid tumors.

DETAILED DESCRIPTION:
The study consists of 2 parts, a dose-escalation part (Phase 1) and an expansion part (Phase 2). Both parts will enroll participants with advanced non-resectable NSCLC, advanced non-resectable thyroid cancer and other advanced solid tumors that have progressed following standard systemic therapy, have not adequately responded to standard systemic therapy, or the participants must be intolerant to or the Investigator has determined that treatment with standard therapy is not appropriate, or there must be no accepted standard therapy for their disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis during dose escalation (Phase 1) - Pathologically documented, definitively diagnosed non-resectable advanced solid tumor.

  * All participants treated at doses > 120 mg per day must have MTC, or a RET-altered solid tumor per local assessment of tumor tissue and/or blood.
* Diagnosis during dose expansion (Phase 2) - All participants (with the exception of participants with MTC enrolled in Groups 3, 4, and 9) must have an oncogenic RET-rearrangement/fusion or mutation (excluding synonymous, frameshift, and nonsense mutations) solid tumor, as determined by local or central testing of tumor or circulating tumor nucleic acid in blood; as detailed below.

  * Group 1 - participants must have pathologically documented, definitively diagnosed locally advanced or metastatic NSCLC with a RET fusion previously treated with a platinum-based chemotherapy.
  * Group 2 - participants must have pathologically documented, definitively diagnosed locally advanced or metastatic NSCLC with a RET fusion not previously treated with a platinum-based chemotherapy, including those who have not had any systemic therapy. Prior platinum chemotherapy in the neoadjuvant and adjuvant setting is permitted if the last dose of platinum was 4 months or more before the first dose of study drug.
  * Group 3 - participants must have pathologically documented, definitively diagnosed advanced MTC that had progressed within 14 months prior to the Screening Visit and was previously treated with cabozantinib and/or vandetanib.
  * Group 4 - participants must have pathologically documented, definitively diagnosed advanced MTC that had progressed within 14 months prior to the Screening Visit and was not previously treated with cabozantinib and/or vandetanib.
  * Group 5 - participants must have a pathologically documented, definitively diagnosed advanced solid tumor with an oncogenic RET fusion, have previously received standard of care (SOC) appropriate for their tumor type (unless there is no accepted standard therapy for the tumor type or the Investigator has determined that treatment with standard therapy is not appropriate), and must not have been eligible for any of the other groups.
  * Group 6 - participants must have a pathologically documented, definitively diagnosed advanced solid tumor with an oncogenic RET fusion or mutation that was previously treated with a selective tyrosine kinase inhibitor (TKI) that inhibits RET
  * Group 7 - participants must have a pathologically documented, definitively diagnosed advanced solid tumor with an oncogenic RET mutation previously treated with SOC appropriate for the tumor type and not eligible for any of the other groups
  * Group 8 - participants must have pathologically documented, definitively diagnosed locally advanced or metastatic NSCLC with a RET fusion that was previously treated with a platinum based chemotherapy (China only).
  * Group 9 - participants must have pathologically documented, definitively diagnosed advanced MTC that had progressed within 14 months prior to the Screening Visit, and was not previously treated with systemic therapy (except prior cytotoxic chemotherapy is allowed) for advanced or metastatic disease (China only).
* Participants must have non-resectable disease.
* Dose expansion (Phase 2): Participants in all groups (except Group 7) must have measurable disease per RECIST v1.1 (or RANO, criteria if appropriate for tumor type).
* Participants agrees to provide tumor tissue (archived, if available or a fresh biopsy) for RET status confirmation and is willing to consider an on-treatment tumor biopsy, if considered safe and medically feasible by the treating Investigator. For Phase 2, Group 6, participants are required to undergo a pretreatment biopsy to define baseline RET status in tumor tissue.
* Participants has Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.

Key Exclusion Criteria:

* Participant's cancer has a known primary driver alteration other than RET. For example, NSCLC with a targetable mutation in EGFR, ALK, ROS1 or BRAF; colorectal with an oncogenic KRAS, NRAS, or BRAF mutation.
* Participants had any of the following within 14 days prior to the first dose of study drug:

  1. Platelet count < 75 × 10^9/L.
  2. Absolute neutrophil count < 1.0 × 10^9/L.
  3. Hemoglobin < 9.0 g/dL (red blood cell transfusion and erythropoietin may be used to reach at least 9.0 g/dL, but must have been administered at least 2 weeks prior to the first dose of study drug.
  4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 × the upper limit of normal (ULN) if no hepatic metastases are present; > 5 × ULN if hepatic metastases are present.
  5. Total bilirubin > 1.5 × ULN; > 3 × ULN with direct bilirubin > 1.5 × ULN in presence of Gilbert's disease.
  6. Estimated (Cockcroft-Gault formula) or measured creatinine clearance < 40 mL/min.
  7. Total serum phosphorus > 5.5 mg/dL
* QT interval corrected using Fridericia's formula (QTcF) > 470 msec or history of prolonged QT syndrome or Torsades de pointes, or familial history of prolonged QT syndrome.
* Clinically significant, uncontrolled, cardiovascular disease.
* Central nervous system (CNS) metastases or a primary CNS tumor that is associated with progressive neurological symptoms.
* Clinically symptomatic interstitial lung disease or interstitial pneumonitis including radiation pneumonitis
* Participants in Groups 1-5 and 7 (Phase 2) previously treated with a selective RET inhibitor
* Participant had a major surgical procedure within 14 days of the first dose of study drug
* Participant had a history of another primary malignancy that had been diagnosed or required therapy within the a year prior to the study
* Pregnant or breastfeeding female participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (69):
- United States (18):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - UC Irvine Medical Center, Orange, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Massachusetts General Hospital., Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Antwerp University Hospital, Edegem, Belgium
- China (15):
  - Beijing Cancer Hospital, Beijing
  - The affiliated Cancer Hospital, School of Medicine, UESTC, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - Fujian Provincial Cancer Hospital, Fuzhou
  - First Affiliated Hospital of Gannan Medical University, Ganzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Guangdong General Hospital, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Jinan Central Hospital, Jinan
  - Gansu Cancer Hospital, Lanzhou
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjing
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital, Zhengzhou
- France (8):
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier Régional Universitaire de Lille (CHRU) - Hôpital Claude Huriez, Lille
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - CHU de Rennes - Hopital de Pontchaillo, Rennes
  - Hôpital Larrey, Toulouse
  - Gustave Roussy, Villejuif
- Germany (5):
  - Helios Klinikum Emil von Behring GmbH, Berlin
  - Universitätsklinikum Essen, Essen
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Klinikum der Universität München, München
  - Pius-Hospital, Oldenburg
- The Chinese University of Hong Kong, Shatin, Hong Kong
- Italy (4):
  - Ospedale Santa Maria Delle Croci, Ravenna, Emilia-Romagna
  - Istituto Nazionale Tumori Regina Elena, Rome, Lazio
  - IEO, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
- Netherlands (2):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
- National Cancer Centre, Singapore, Singapore
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (5):
  - Institut Catala d Oncologia Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (3):
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Subbiah V, Hu MI, Mansfield AS, Taylor MH, Schuler M, Zhu VW, Hadoux J, Curigliano G, Wirth L, Gainor JF, Alonso G, Adkins D, Godbert Y, Ahn MJ, Cassier PA, Cho BC, Lin CC, Zalutskaya A, Barata T, Trask P, Scalori A, Bordogna W, Heinzmann S, Brose MS. Pralsetinib in Patients with Advanced/Metastatic Rearranged During Transfection (RET)-Altered Thyroid Cancer: Updated Efficacy and Safety Data from the ARROW Study. Thyroid. 2024 Jan;34(1):26-40. doi: 10.1089/thy.2023.0363. PMID 38009200
- [Derived] Subbiah V, Burris HA 3rd, Kurzrock R. Revolutionizing cancer drug development: Harnessing the potential of basket trials. Cancer. 2024 Jan;130(2):186-200. doi: 10.1002/cncr.35085. Epub 2023 Nov 7. PMID 37934000
- [Derived] Griesinger F, Curigliano G, Subbiah V, Baik CS, Tan DS, Lee DH, Misch D, Garralda E, Kim DW, van der Wekken AJ, Gainor JF, Paz-Ares L, Liu SV, Kalemkerian GP, Bowles DW, Mansfield AS, Lin JJ, Smoljanovic V, Rahman A, Zalutskaya A, Louie-Gao M, Boral AL, Mazieres J. Pralsetinib in patients with RET fusion-positive non-small-cell lung cancer: A plain language summary of the ARROW study. Future Oncol. 2024 Feb;20(6):297-306. doi: 10.2217/fon-2023-0155. Epub 2023 Nov 2. PMID 37916501
- [Derived] Zhou Q, Zhao J, Chang J, Wang H, Fan Y, Wang K, Wu G, Nian W, Sun Y, Sun M, Wang X, Shi H, Zheng X, Yao S, Qin M, Shen Z, Yang J, Wu YL. Efficacy and safety of pralsetinib in patients with advanced RET fusion-positive non-small cell lung cancer. Cancer. 2023 Oct 15;129(20):3239-3251. doi: 10.1002/cncr.34897. Epub 2023 Jun 6. PMID 37282666
- [Derived] Subbiah V, Cassier PA, Siena S, Garralda E, Paz-Ares L, Garrido P, Nadal E, Vuky J, Lopes G, Kalemkerian GP, Bowles DW, Seetharam M, Chang J, Zhang H, Green J, Zalutskaya A, Schuler M, Fan Y, Curigliano G. Pan-cancer efficacy of pralsetinib in patients with RET fusion-positive solid tumors from the phase 1/2 ARROW trial. Nat Med. 2022 Aug;28(8):1640-1645. doi: 10.1038/s41591-022-01931-y. Epub 2022 Aug 12. PMID 35962206
- [Derived] Popat S, Liu SV, Scheuer N, Hsu GG, Lockhart A, Ramagopalan SV, Griesinger F, Subbiah V. Addressing challenges with real-world synthetic control arms to demonstrate the comparative effectiveness of Pralsetinib in non-small cell lung cancer. Nat Commun. 2022 Jun 17;13(1):3500. doi: 10.1038/s41467-022-30908-1. PMID 35715405
- [Derived] Subbiah V, Hu MI, Wirth LJ, Schuler M, Mansfield AS, Curigliano G, Brose MS, Zhu VW, Leboulleux S, Bowles DW, Baik CS, Adkins D, Keam B, Matos I, Garralda E, Gainor JF, Lopes G, Lin CC, Godbert Y, Sarker D, Miller SG, Clifford C, Zhang H, Turner CD, Taylor MH. Pralsetinib for patients with advanced or metastatic RET-altered thyroid cancer (ARROW): a multi-cohort, open-label, registrational, phase 1/2 study. Lancet Diabetes Endocrinol. 2021 Aug;9(8):491-501. doi: 10.1016/S2213-8587(21)00120-0. Epub 2021 Jun 9. PMID 34118198
- [Derived] Gainor JF, Curigliano G, Kim DW, Lee DH, Besse B, Baik CS, Doebele RC, Cassier PA, Lopes G, Tan DSW, Garralda E, Paz-Ares LG, Cho BC, Gadgeel SM, Thomas M, Liu SV, Taylor MH, Mansfield AS, Zhu VW, Clifford C, Zhang H, Palmer M, Green J, Turner CD, Subbiah V. Pralsetinib for RET fusion-positive non-small-cell lung cancer (ARROW): a multi-cohort, open-label, phase 1/2 study. Lancet Oncol. 2021 Jul;22(7):959-969. doi: 10.1016/S1470-2045(21)00247-3. Epub 2021 Jun 9. PMID 34118197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 590 participants with rearranged during transfection (RET) fusion-positive non-small cell lung cancer (NSCLC), RET mutation-positive medullary thyroid cancer (also known as RET-mutant MTC), RET fusion-positive thyroid cancer (TC) and other advanced solid tumors took part in the study at 74 investigative sites across 13 countries from 17 March 2017 to 21 March 2024. The study was divided into two parts: Phase 1 (Dose Escalation) and Phase 2 (Dose Expansion).
Pre-assignment Details: For Phase I, The number of participants in each arm within the participant flow reflects the arms they were originally assigned to, whereas numbers reported in the pharmacokinetics outcome measure (OM) represent the number based on actual treatment received by the participants. 1 participant assigned to the 200/100 mg arm received the 100/100 mg treatment. Hence, was counted under the 100/100 mg arm in the PK-evaluable population.
Groups:
- Phase I: Pralsetinib 30 mg: Participants received pralsetinib 30 milligrams (mg), orally, once a day (QD) until discontinuation due to toxicity, disease progression, or other reasons.
- Phase I: Pralsetinib 60 mg: Participants received pralsetinib 60 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- Phase I: Pralsetinib 100 mg: Participants received pralsetinib 100 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- Phase I: Pralsetinib 200 mg: Participants received pralsetinib 200 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- Phase I: Pralsetinib 300 mg: Participants received pralsetinib 300 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- Phase I: Pralsetinib 400 mg: Participants received pralsetinib 400 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- Phase I: Pralsetinib 600 mg: Participants received pralsetinib 600 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- Phase I: Pralsetinib 100/100 mg: Participants received pralsetinib 100 mg, orally, twice a day (BID) until discontinuation due to toxicity, disease progression, or other reasons.
- Phase I: Pralsetinib 200/100 mg: Participants received pralsetinib 200 mg in the morning and then 100 mg in the evening orally until discontinuation due to toxicity, disease progression, or other reasons.
- Phase II: Pralsetinib 400 mg: Participants with advanced NSCLC, advanced non-resectable TC and other advanced non-resectable solid tumors with various rearranged during transfection (RET)-alterations were enrolled in this arm to receive pralsetinib, 400 mg, QD until discontinuation due to toxicity, disease progression, or other reasons.
Period: Overall Study
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg | Phase II: Pralsetinib 400 mg
Started | 2 | 6 | 5 | 13 | 11 | 12 | 4 | 5 | 4 | 528
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 6 | 5 | 13 | 11 | 12 | 4 | 5 | 4 | 528
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Death | 1 | 4 | 2 | 2 | 5 | 2 | 1 | 4 | 3 | 240
Not completed — Initiation of Another Therapy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 16
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 1 | 1 | 5 | 2 | 0 | 1 | 0 | 0 | 30
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 52
Not completed — Reason Not Specified | 0 | 1 | 0 | 4 | 3 | 6 | 2 | 0 | 1 | 181

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who had received at least 1 dose of the study drug regardless of the starting dose levels.
Groups:
- Phase I: Pralsetinib 30 mg: Participants received pralsetinib 30 milligrams (mg) orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- Total: Total of all reporting groups
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg | Phase II: Pralsetinib 400 mg | Total
Number analyzed (Participants) | 2 | 6 | 5 | 13 | 11 | 12 | 4 | 5 | 4 | 528 | 590
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (9.2) | 49.5 (18.0) | 51.2 (13.2) | 53.8 (13.6) | 60.6 (11.0) | 49.2 (17.8) | 59.5 (9.1) | 63.0 (11.09) | 61.8 (18.25) | 57.7 (12.6) | 57.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 5 | 4 | 3 | 3 | 1 | 2 | 257 | 283
  Male | 1 | 3 | 1 | 8 | 7 | 9 | 1 | 4 | 2 | 271 | 307
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 19 | 28
  Not Hispanic or Latino | 0 | 4 | 4 | 12 | 11 | 9 | 4 | 3 | 4 | 465 | 516
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 44 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 203 | 209
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 6
  White | 0 | 3 | 2 | 11 | 11 | 9 | 4 | 3 | 4 | 284 | 331
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Unknown or Not Reported | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 32 | 39

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 : Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of Pralsetinib
Description: MTD was defined as the highest tolerated dose of pralsetinib without causing dose limiting toxicities (DLTs). DLT was defined as any Grade ≥3 adverse event (AE) occurring during Cycle 1 during Phase 1 (dose escalation) that is not clearly caused by something other than pralsetinib. RP2D was defined as the highest dose with acceptable toxicity as determined from dose-escalation phase.
Time Frame: Up to approximately 30.8 months
Population: Dose-determining population included all participants in the dose-escalation part who have received ≥75% (21 days) of the study drug and completed safety evaluations through Cycle 1 Day 28 or experienced a DLT.
Measure: Number; unit: mg
Groups:
- Phase 1: All Participants QD: Participants received pralsetinib at varying doses at a QD schedule until discontinuation due to toxicity, disease progression, or other reasons.
Arm/Group | Phase 1: All Participants QD
Number analyzed (Participants) | 51
mg
  MTD | 400
  RP2D | 400

2. Primary Outcome: Phase 1 and Phase 2: Number of Participants With AEs and Serious AEs (SAEs)
Description: An AE was any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. A SAE is any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: From Cycle 1 Day 1 up to 30 days after the final dose of study drug (up to approximately 6.7 years)
Population: Safety Population included all participants who have received at least 1 dose of the study drug regardless of starting dose levels. As pre-specified in the SAP, safety data was to be analyzed and reported as per the pre-planned grouped dose level II (SAP section 3.6.5.2). Hence, per dose safety data is not presented for this study.
Measure: Number; unit: percentage of participants
Groups:
- Pralsetinib ≤ 300 mg QD: Participants received pralsetinib, 300 mg or less, orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- Pralsetinib 400 mg QD: Participants received pralsetinib, 400 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- Pralsetinib BID Dosing Schedule: Participants received pralsetinib, 100 mg, orally, BID or 200 mg in the morning and then 100 mg in the evening, orally, until discontinuation due to toxicity, disease progression, or other reasons.
- Pralsetinib All Doses: Participants received pralsetinib at varying doses at the QD and BID schedule until discontinuation due to toxicity, disease progression, or other reasons.
Arm/Group | Pralsetinib ≤ 300 mg QD | Pralsetinib 400 mg QD | Pralsetinib BID Dosing Schedule | Pralsetinib All Doses
Number analyzed (Participants) | 37 | 540 | 9 | 590
percentage of participants
  AEs | 37 | 540 | 9 | 590
  SAEs | 26 | 381 | 7 | 416

3. Primary Outcome: Phase 2: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) for at least two assessments with at least 28 days apart and no disease progression (PD) in between. Per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1), CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in the short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters (SOD) of all target lesions, taking as reference the baseline SOD, in the absence of CR. PD was defined as at least a 20% increase in SOD of target lesions, taking as reference the smallest SOD on study (including baseline). ORR and its two-sided 95% CI, based on the exact binomial distribution (Clopper-Pearson), were presented.
Time Frame: Up to approximately 79.8 months
Population: RET-altered measurable disease population included participants in the efficacy population who had measurable (target) disease per RECIST v1.1 at baseline according to blinded central review (BICR) and sufficient evidence of a RET alteration. As prespecified in the SAP, Phase 1 participants treated at 400 mg QD are also included in Phase 2 efficacy analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- RET- Fusion Positive NSCLC With Prior Platinum Treatment:: Participants who had RET-fusion positive NSCLC previously treated with platinum-based chemotherapies received pralsetinib, 400 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- RET-fusion Positive NSCLC With Non-platinum Systemic Treatment: Participants who had RET-fusion positive NSCLC previously treated with non-platinum or systemic therapies received pralsetinib, 400 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment: Participants who had RET-fusion positive NSCLC not previously treated with systemic or platinum-based chemotherapies received pralsetinib, 400 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- RET-mutation MTC With Prior Cabozantinib and/or Vandetanib Treatment: Participants who had RET- mutation positive MTC previously treated with either cabozantinib and/or vandetanib therapies received pralsetinib, 400 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- RET-mutation MTC With No Prior Cabozantinib or Vandetanib Treatment: Participants who had RET- mutation positive MTC not previously treated with cabozantinib or vandetanib therapies received pralsetinib, 400 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- RET-fusion Positive TC: Participants who had RET-fusion positive TC received pralsetinib, 400 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- RET-fusion Positive Solid Tumors Other Than NSCLC and TC: Participants who had other RET-positive solid tumors other than NSCLC and TC received pralsetinib, 400 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- RET-altered Solid Tumors Previously Treated With RET Inhibitor: Participants who had RET-altered (fusion or mutation) solid tumors previously treated with a selective RET tyrosine kinase inhibitor (TKI) received pralsetinib, 400 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- RET-mutation Positive Tumors Other Than MTC: Participants who had RET-mutation positive solid tumors received pralsetinib, 400 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment: | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment | RET-mutation MTC With Prior Cabozantinib and/or Vandetanib Treatment | RET-mutation MTC With No Prior Cabozantinib or Vandetanib Treatment | RET-fusion Positive TC | RET-fusion Positive Solid Tumors Other Than NSCLC and TC | RET-altered Solid Tumors Previously Treated With RET Inhibitor | RET-mutation Positive Tumors Other Than MTC
Number analyzed (Participants) | 130 | 23 | 106 | 60 | 72 | 27 | 28 | 21 | 13
percentage of participants | 63.1 [54.2 to 71.4] | 73.9 [51.6 to 89.8] | 78.3 [69.2 to 85.7] | 56.7 [43.2 to 69.4] | 77.8 [66.4 to 86.7] | 85.2 [66.3 to 95.8] | 46.4 [27.5 to 66.1] | 19.0 [5.4 to 41.9] | 7.7 [0.99 to 36.0]

4. Secondary Outcome: Phase 1: ORR
Description: ORR was defined as the percentage of participants with a confirmed CR or PR for at least two assessments with at least 28 days apart and no PD in between. Per RECIST v1.1, CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in the short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. PD was defined as at least a 20% increase in SOD of target lesions, taking as reference the smallest SOD on study (including baseline). ORR and its two-sided 95% CI, based on the exact binomial distribution (Clopper-Pearson), was presented.
Time Frame: Up to approximately 28 months
Population: Efficacy population included all participants who have been exposed to at least one dose of the study drug on or prior to 11 July 2019.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase I: Pralsetinib 30 mg: Participants received pralsetinib 30 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- Phase I: Pralsetinib 200 mg: Participants received pralsetinib 200 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- Phase I: Pralsetinib 400 mg: Participants received pralsetinib 400 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- Phase I: Pralsetinib 600 mg: Participants received pralsetinib 600 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
- Phase I: Pralsetinib 100/100 mg: Participants received pralsetinib 100 mg, orally, BID until discontinuation due to toxicity, disease progression, or other reasons.
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg
Number analyzed (Participants) | 2 | 6 | 5 | 13 | 11 | 12 | 4 | 5 | 4
percentage of participants | 0 [NA to NA] — The 95% confidence interval (CI) was not estimable due to insufficient number of participants with events. | 50.0 [11.8 to 88.2] | 40.0 [5.3 to 85.3] | 38.5 [13.9 to 68.4] | 45.5 [16.7 to 76.6] | 41.7 [15.2 to 72.3] | 25.0 [0.99 to 80.6] | 80.0 [28.4 to 99.5] | 75.0 [19.4 to 99.4]

5. Secondary Outcome: Phase 1 and Phase 2: ORR in RET-fusion Positive NSCLC Participants With Specific RET Gene Status
Description: Oncogenic RET rearrangements have been identified in 1%-2% of NSCLC. These rearrangements typically produce chimeric transcripts that encode a fusion protein consisting of the RET kinase domain coupled to a protein with a dimerization domain (e.g., Kinesin family member 5B (KIF5B), coiled-coil domain containing 6 (CCDC6), nuclear receptor coactivator 4 (NCOA4)). RET genotypes were determined by local testing and/or central analysis of circulating tumor deoxyribonucleic acid (ctDNA). ORR was assessed in participants having specific RET rearrangements. ORR was defined as the percentage of participants with a confirmed CR or PR for at least 2 assessments with at least 28 days apart and no PD in between. CR, PR, and PD were defined per RECIST as outlined in the description for OM 3.
Time Frame: Up to approximately 79.8 months
Population: RET-altered measurable disease population included participants in the efficacy population who have measurable (target) disease per RECIST v1.1, at baseline according to BICR and sufficient evidence of a RET alteration. As prespecified in the SAP, Phase 1 participants treated at 400 mg QD are pooled with Phase 2 participants for efficacy analysis. Number analyzed is the number of participants with the specified mutation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- RET- Fusion Positive NSCLC With Prior Platinum Treatment: Participants who had RET-fusion positive NSCLC previously treated with platinum-based chemotherapies received pralsetinib, 400 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment
Number analyzed (Participants) | 130 | 23 | 106
percentage of participants
  KIF5B: number analyzed (Participants) | 91 | 17 | 76
  KIF5B | 63.7 [53.0 to 73.6] | 82.4 [56.6 to 96.2] | 78.9 [68.1 to 87.5]
  CCDC6: number analyzed (Participants) | 25 | 4 | 19
  CCDC6 | 68.0 [46.5 to 85.1] | 75.0 [19.4 to 99.4] | 84.2 [60.4 to 96.6]
  NCOA4: number analyzed (Participants) | 1 | 0 | 0
  NCOA4 | 100 [2.5 to 100] |  |
  Other: number analyzed (Participants) | 13 | 2 | 11
  Other | 46.2 [19.2 to 74.9] | 0 [NA to NA] — The 95% CI was not estimable due to insufficient number of participants with events. | 63.6 [30.8 to 89.1]

6. Secondary Outcome: Phase 1 and Phase 2: ORR in RET-mutation MTC Participants With Specific RET Gene Status
Description: Oncogenic RET activation has been implicated as a driver in MTC. These rearrangements typically produce chimeric transcripts that encode a fusion protein consisting of the RET kinase domain coupled to a protein with a dimerization domain (e.g., M918T, cysteine rich domain, V804X). RET genotypes were determined by local testing and/or central analysis of ctDNA. ORR was assessed in participants having specific RET rearrangements. ORR was defined as the percentage of participants with a confirmed CR or PR for at least 2 assessments with at least 28 days apart and no PD in between. CR, PR, and PD were defined per RECIST as outlined in the description for OM 3.
Time Frame: Up to approximately 79.8 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RET-mutation MTC With Prior Cabozantinib and/or Vandetanib Treatment | RET-mutation MTC With No Prior Cabozantinib or Vandetanib Treatment
Number analyzed (Participants) | 60 | 72
percentage of participants
  M918T: number analyzed (Participants) | 41 | 43
  M918T | 53.7 [37.4 to 69.3] | 74.4 [58.8 to 86.5]
  Cysteine Rich Domain: number analyzed (Participants) | 13 | 25
  Cysteine Rich Domain | 46.2 [19.2 to 74.9] | 88.0 [68.8 to 97.5]
  V804X: number analyzed (Participants) | 2 | 1
  V804X | 100 [15.8 to 100] | 0 [NA to NA] — Since only 1 participant was analyzed upper and lower limit of 95% CI was not evaluable.
  Other: number analyzed (Participants) | 4 | 3
  Other | 100 [39.8 to 100] | 66.7 [9.4 to 99.2]

7. Secondary Outcome: Phase 1 and Phase 2: ORR in RET-fusion Positive TC Participants With Specific RET Gene Status
Description: Oncogenic RET activation has been implicated as a driver in both MTC and differentiated TC (DTC). These rearrangements typically produce chimeric transcripts that encode a fusion protein consisting of the RET kinase domain coupled to a protein with a dimerization domain (e.g., KIF5B, CCDC6, NCOA4). RET genotypes were determined by local testing and/or central analysis of ctDNA. ORR was assessed in participants having specific RET rearrangements. ORR was defined as the percentage of participants with a confirmed CR or PR for at least 2 assessments with at least 28 days apart and no PD in between. CR, PR, and PD were defined per RECIST as outlined in the description for OM 3.
Time Frame: Up to approximately 79.8 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- RET-fusion Positive TC: Participants who had RET-fusion positive TC received pralsetinib 400 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
Arm/Group | RET-fusion Positive TC
Number analyzed (Participants) | 27
percentage of participants
  KIF5B: number analyzed (Participants) | 0
  CCDC6: number analyzed (Participants) | 17
  CCDC6 | 82.4 [56.6 to 96.2]
  NCOA4: number analyzed (Participants) | 6
  NCOA4 | 100 [54.1 to 100]
  Other: number analyzed (Participants) | 4
  Other | 75.0 [19.4 to 99.4]

8. Secondary Outcome: Phase 1 and Phase 2: Clinical Benefit Rate (CBR) in RET-fusion Positive NSCLC Participants With Specific RET Gene Status
Description: Oncogenic RET rearrangements have been identified in 1%-2% of NSCLC. These rearrangements typically produce chimeric transcripts that encode a fusion protein consisting of the RET kinase domain coupled to a protein with a dimerization domain (e.g., KIF5B, CCDC6, NCOA4). RET genotypes were determined by local testing and/or central analysis of ctDNA. CBR was assessed in participants having specific RET rearrangements. CBR was defined as the percentage of participants with a confirmed CR or PR, or stable disease (SD) which has been lasting at least 16 weeks (i.e. 4 cycles if 28 days are in one cycle) from the first dose date. CR and PR were defined per RECIST as outlined in the description for OM 3. SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in SOD of target lesions, taking as reference the smallest SOD on study (including baseline).
Time Frame: Up to approximately 79.8 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment
Number analyzed (Participants) | 130 | 23 | 106
percentage of participants
  KIF5B: number analyzed (Participants) | 91 | 17 | 76
  KIF5B | 76.9 [66.9 to 85.1] | 88.2 [63.6 to 98.5] | 81.6 [71.0 to 89.5]
  CCDC6: number analyzed (Participants) | 25 | 4 | 19
  CCDC6 | 76.0 [54.9 to 90.6] | 75.0 [19.4 to 99.4] | 84.2 [60.4 to 96.6]
  NCOA4: number analyzed (Participants) | 1 | 0 | 0
  NCOA4 | 100 [2.5 to 100] |  |
  Other: number analyzed (Participants) | 13 | 2 | 11
  Other | 53.8 [25.1 to 80.8] | 0 [NA to NA] — The 95% CI was not estimable due to insufficient number of participants with events. | 63.6 [30.8 to 89.1]

9. Secondary Outcome: Phase 1 and Phase 2: CBR in RET-mutation MTC Participants With Specific RET Gene Status
Description: Oncogenic RET activation has been implicated as a driver in MTC. These rearrangements typically produce chimeric transcripts that encode a fusion protein consisting of the RET kinase domain coupled to a protein with a dimerization domain (e.g., M918T, cysteine rich domain, V804X). RET genotypes were determined by local testing and/or central analysis of ctDNA. CBR was assessed in participants having specific RET rearrangements. CBR was defined as the percentage of participants with a confirmed CR or PR, or SD which has been lasting at least 16 weeks (i.e. 4 cycles if 28 days are in one cycle) from the first dose date. CR and PR were defined per RECIST as outlined in the description for OM 3. SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in SOD of target lesions, taking as reference the smallest SOD on study (including baseline).
Time Frame: Up to approximately 79.8 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RET-mutation MTC With Prior Cabozantinib and/or Vandetanib Treatment | RET-mutation MTC With No Prior Cabozantinib or Vandetanib Treatment
Number analyzed (Participants) | 60 | 72
percentage of participants
  M918T: number analyzed (Participants) | 41 | 43
  M918T | 78.0 [62.4 to 89.4] | 86.0 [72.1 to 94.7]
  Cysteine Rich Domain: number analyzed (Participants) | 13 | 25
  Cysteine Rich Domain | 76.9 [46.2 to 95.0] | 96.0 [79.6 to 99.9]
  V804X: number analyzed (Participants) | 2 | 1
  V804X | 100 [15.8 to 100] | 100 [2.5 to 100]
  Other: number analyzed (Participants) | 4 | 3
  Other | 100 [39.8 to 100] | 100 [29.2 to 100]

10. Secondary Outcome: Phase 1 and Phase 2: CBR in RET-fusion Positive TC Participants With Specific RET Gene Status
Description: Oncogenic RET activation has been implicated as a driver in both MTC and DTC. These rearrangements typically produce chimeric transcripts that encode a fusion protein consisting of the RET kinase domain coupled to a protein with a dimerization domain (e.g., KIF5B, CCDC6, NCOA4). RET genotypes were determined by local testing and/or central analysis of ctDNA. CBR was assessed in participants having specific RET rearrangements. CBR was defined as the percentage of participants with a confirmed CR or PR or SD which has been lasting at least 16 weeks (i.e. 4 cycles if 28 days are in one cycle) from the first dose date. CR and PR were defined per RECIST as outlined in the description for OM 3. SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in SOD of target lesions, taking as reference the smallest SOD on study (including baseline).
Time Frame: Up to approximately 79.8 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RET-fusion Positive TC
Number analyzed (Participants) | 27
percentage of participants
  KIF5B: number analyzed (Participants) | 0
  CCDC6: number analyzed (Participants) | 17
  CCDC6 | 82.4 [56.6 to 96.2]
  NCOA4: number analyzed (Participants) | 6
  NCOA4 | 100 [54.1 to 100]
  Other: number analyzed (Participants) | 4
  Other | 75.0 [19.4 to 99.4]

11. Secondary Outcome: Phase 1 and Phase 2: Disease Control Rate (DCR) in RET-fusion Positive NSCLC Participants With Specific RET Gene Status
Description: Oncogenic RET rearrangements have been identified in 1%-2% of NSCLC. These rearrangements typically produce chimeric transcripts that encode a fusion protein consisting of the RET kinase domain coupled to a protein with a dimerization domain (e.g., KIF5B, CCDC6, NCOA4). RET genotypes were determined by local testing and/or central analysis of ctDNA. DCR was assessed in participants having specific RET rearrangements. DCR was defined as the percentage of participants with a confirmed CR/PR, or SD. CR and PR were defined per RECIST as outlined in the description for OM 3. SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in SOD of target lesions, taking as reference the smallest SOD on study (including baseline).
Time Frame: Up to approximately 79.8 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment
Number analyzed (Participants) | 130 | 23 | 106
percentage of participants
  KIF5B: number analyzed (Participants) | 91 | 17 | 76
  KIF5B | 93.4 [86.2 to 97.5] | 94.1 [71.3 to 99.9] | 88.2 [78.7 to 94.4]
  CCDC6: number analyzed (Participants) | 25 | 4 | 19
  CCDC6 | 88.0 [68.8 to 97.5] | 100 [39.8 to 100] | 89.5 [66.9 to 98.7]
  NCOA4: number analyzed (Participants) | 1 | 0 | 0
  NCOA4 | 100 [2.5 to 100] |  |
  Other: number analyzed (Participants) | 13 | 2 | 11
  Other | 84.6 [54.6 to 98.1] | 50.0 [1.3 to 98.7] | 100 [71.5 to 100]

12. Secondary Outcome: Phase 1 and Phase 2: DCR in RET-mutation MTC Participants With Specific RET Gene Status
Description: Oncogenic RET activation has been implicated as a driver in MTC. These rearrangements typically produce chimeric transcripts that encode a fusion protein consisting of the RET kinase domain coupled to a protein with a dimerization domain (e.g., M918T, cysteine rich domain, V804X). RET genotypes were determined by local testing and/or central analysis of ctDNA. DCR was assessed in participants having specific RET rearrangements. DCR was defined as the percentage of participants with a confirmed CR/PR, or SD. CR and PR were defined per RECIST as outlined in the description for OM 3. SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in SOD of target lesions, taking as reference the smallest SOD on study (including baseline).
Time Frame: Up to approximately 79.8 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RET-mutation MTC With Prior Cabozantinib and/or Vandetanib Treatment | RET-mutation MTC With No Prior Cabozantinib or Vandetanib Treatment
Number analyzed (Participants) | 60 | 72
percentage of participants
  M918T: number analyzed (Participants) | 41 | 43
  M918T | 95.1 [83.5 to 99.4] | 90.7 [77.9 to 97.4]
  Cysteine Rich Domain: number analyzed (Participants) | 13 | 25
  Cysteine Rich Domain | 92.3 [64.0 to 99.8] | 96.0 [79.6 to 99.9]
  V804X: number analyzed (Participants) | 2 | 1
  V804X | 100 [15.8 to 100] | 100 [2.5 to 100]
  Other: number analyzed (Participants) | 4 | 3
  Other | 100 [39.8 to 100] | 100 [29.2 to 100]

13. Secondary Outcome: Phase 1 and Phase 2: DCR in RET-fusion Positive TC Participants With Specific RET Gene Status
Description: Oncogenic RET activation has been implicated as a driver in both MTC and DTC. These rearrangements typically produce chimeric transcripts that encode a fusion protein consisting of the RET kinase domain coupled to a protein with a dimerization domain (e.g., KIF5B, CCDC6, NCOA4). RET genotypes were determined by local testing and/or central analysis of ctDNA. DCR was assessed in participants having specific RET rearrangements. DCR was defined as the percentage of participants with a confirmed CR/PR, or SD. CR and PR were defined per RECIST as outlined in the description for OM 3. SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in SOD of target lesions, taking as reference the smallest SOD on study (including baseline).
Time Frame: Up to approximately 79.8 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RET-fusion Positive TC
Number analyzed (Participants) | 27
percentage of participants
  KIF5B: number analyzed (Participants) | 0
  CCDC6: number analyzed (Participants) | 17
  CCDC6 | 94.1 [71.3 to 99.9]
  NCOA4: number analyzed (Participants) | 6
  NCOA4 | 100 [54.1 to 100]
  Other: number analyzed (Participants) | 4
  Other | 100 [39.8 to 100]

14. Secondary Outcome: Phase 1 and Phase 2: Duration of Response (DOR) in RET-mutation NSCLC Participants With Specific RET Gene Status
Description: Oncogenic RET rearrangements have been identified in 1%-2% of NSCLC. These rearrangements typically produce chimeric transcripts that encode a fusion protein consisting of the RET kinase domain coupled to a protein with a dimerization domain (e.g., KIF5), CCDC6, NCOA4). RET genotypes were determined by local testing &/or central analysis of circulating tumor deoxyribonucleic acid (ctDNA). DOR was assessed in participants having specific RET rearrangements. DOR=time from first documented CR/PR to date of first documented PD or death due to any cause, whichever occurs first. Per RECIST, CR=disappearance of all target lesions or any pathological lymph nodes (target or non-target) having a reduction in the short axis to <10 mm. PR=at least a 30% decrease in SOD of all target lesions, taking as reference the baseline SOD, in absence of CR. PD=as at least a 20% increase in SOD of target lesions, taking as reference smallest SOD on study. DOR was analyzed using the Kaplan-Meier (KM) method.
Time Frame: Up to approximately 79.8 months
Population: RET-altered measurable disease population included participants in the efficacy population who have measurable (target) disease per RECIST v1.1, at baseline according to BICR & sufficient evidence of a RET alteration. As prespecified in SAP, Phase 1 participants treated at 400 mg QD are pooled with Phase 2 participants for efficacy analysis. Participants who had a response of CR/PR were analyzed in this outcome measure. Number analyzed is the number of participants with the specified mutation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment
Number analyzed (Participants) | 82 | 17 | 83
months
  KIF5B: number analyzed (Participants) | 58 | 14 | 60
  KIF5B | 15.1 [8.8 to 34.2] | 21.5 [9.3 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 9.2 [7.4 to 13.4]
  CCDC6: number analyzed (Participants) | 17 | 3 | 16
  CCDC6 | 46.7 [33.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 29.6 [11.3 to 47.9] | NA [14.7 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events.
  NCOA4: number analyzed (Participants) | 1 | 0 | 0
  NCOA4 | 12.9 [NA to NA] — The upper and lower limits of 95% CI were not estimable due to insufficient number of participants with events. |  |
  Other: number analyzed (Participants) | 6 | 0 | 7
  Other | 35.2 [10.6 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. |  | 41.2 [27.9 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events.

15. Secondary Outcome: Phase 1 and Phase 2: DOR in RET-mutation MTC Participants With Specific RET Gene Status
Description: Oncogenic RET activation has been implicated as a driver in MTC. These rearrangements typically produce chimeric transcripts that encode a fusion protein consisting of the RET kinase domain coupled to a protein with a dimerization domain (e.g., M918T, cysteine rich domain, V804X). RET genotypes were determined by local testing and/or central analysis of ctDNA. DOR was assessed in participants having specific RET rearrangements. DOR=time from first documented CR/PR to date of first documented PD or death due to any cause, whichever occurs first. Per RECIST, CR= disappearance of all target lesions or any pathological lymph nodes (target or non-target) having a reduction in the short axis to <10 mm. PR=at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in absence of CR. PD=as at least a 20% increase in SOD of target lesions, taking as reference smallest SOD on study (including baseline). DOR was analyzed using the Kaplan-Meier (KM) method.
Time Frame: Up to approximately 79.8 months
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RET-mutation MTC With Prior Cabozantinib and/or Vandetanib Treatment | RET-mutation MTC With No Prior Cabozantinib or Vandetanib Treatment
Number analyzed (Participants) | 34 | 56
months
  M918T: number analyzed (Participants) | 22 | 32
  M918T | 18.4 [15.1 to 25.8] | 51.8 [40.0 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events.
  Cysteine Rich Domain: number analyzed (Participants) | 6 | 22
  Cysteine Rich Domain | 29.5 [8.8 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 36.8 [23.1 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events.
  V804X: number analyzed (Participants) | 2 | 0
  V804X | 21.8 [14.2 to 29.4] |
  Other: number analyzed (Participants) | 4 | 2
  Other | NA [14.5 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — The median and 95% CI was not estimable due to insufficient number of participants with events.

16. Secondary Outcome: Phase 1 and Phase 2: DOR in RET-fusion Positive TC Participants With Specific RET Gene Status
Description: Oncogenic RET activation has been implicated as a driver in MTC. These rearrangements typically produce chimeric transcripts that encode a fusion protein consisting of the RET kinase domain coupled to a protein with a dimerization domain (e.g., KIF5B, CCDC6, NCOA4). RET genotypes were determined by local testing and/or central analysis of ctDNA. DOR was assessed in participants having specific RET rearrangements. DOR=time from first documented CR/PR to date of first documented PD or death due to any cause, whichever occurs first. Per RECIST, CR= disappearance of all target lesions or any pathological lymph nodes (target or non-target) having a reduction in the short axis to <10 mm. PR=at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in absence of CR. PD=as at least a 20% increase in SOD of target lesions, taking as reference smallest SOD on study (including baseline). DOR was analyzed using the KM method.
Time Frame: Up to approximately 79.8 months
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RET-fusion Positive TC
Number analyzed (Participants) | 23
months
  CCDC6: number analyzed (Participants) | 14
  CCDC6 | NA [11.2 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events.
  NCOA4: number analyzed (Participants) | 6
  NCOA4 | 15.2 [6.9 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events.
  Other: number analyzed (Participants) | 3
  Other | NA [23.6 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events.

17. Secondary Outcome: Phase 2: DOR
Description: DOR was defined as the time from first documented response (CR/PR) to the date of first documented PD or death due to any cause, whichever occurs first. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in the short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. PD was defined as at least a 20% increase in SOD of target lesions, taking as reference the smallest SOD on study (including baseline). DOR was analyzed using the KM methods.
Time Frame: Up to approximately 79.8 months
Population: RET-altered measurable disease population included participants in the efficacy population who have measurable (target) disease per RECIST v1.1, at baseline according to BICR & sufficient evidence of a RET alteration. As prespecified in SAP, Phase 1 participants treated at 400 mg QD are pooled with Phase 2 participants for efficacy analysis. Participants who had a response of CR/PR were analyzed in this OM.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- RET-altered Solid Tumors Previously Treated With RET Inhibitor: Participants who had RET-altered (fusion or mutation) solid tumors previously treated with a selective RET TKI received pralsetinib, 400 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons.
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment | RET-mutation MTC With Prior Cabozantinib and/or Vandetanib Treatment | RET-mutation MTC With No Prior Cabozantinib or Vandetanib Treatment | RET-fusion Positive TC | RET-fusion Positive Solid Tumors Other Than NSCLC and TC | RET-altered Solid Tumors Previously Treated With RET Inhibitor | RET-mutation Positive Tumors Other Than MTC
Number analyzed (Participants) | 82 | 17 | 83 | 34 | 56 | 23 | 13 | 4 | 1
months | 31.8 [15.1 to 40.4] | 22.6 [11.1 to 47.9] | 13.4 [9.4 to 21.7] | 21.7 [15.1 to 34.8] | 51.8 [36.8 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [12.9 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 11.1 [5.5 to 25.1] | NA [6.0 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 5.5 [NA to NA] — The 95% CI was not estimable due to insufficient number of participants with events.

18. Secondary Outcome: Phase 2: CBR
Description: CBR was defined as the percentage of participants with CR or PR, or SD which has been lasting at least 16 weeks (i.e. 4 cycles if 28 days are in one cycle) from the first dose date. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in the short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in SOD of target lesions, taking as reference the smallest SOD on study (including baseline). CBR and its two-sided 95% CI, which is based on the exact binomial distribution (Clopper-Pearson), were presented.
Time Frame: Up to approximately 79.8 months
Population: RET-altered measurable disease population included participants in the efficacy population who have measurable (target) disease per RECIST v1.1, at baseline according to BICR and sufficient evidence of a RET alteration. As prespecified in the SAP, Phase 1 participants treated at 400 mg QD are pooled with Phase 2 participants for efficacy analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment | RET-mutation MTC With Prior Cabozantinib and/or Vandetanib Treatment | RET-mutation MTC With No Prior Cabozantinib or Vandetanib Treatment | RET-fusion Positive TC | RET-fusion Positive Solid Tumors Other Than NSCLC and TC | RET-altered Solid Tumors Previously Treated With RET Inhibitor | RET-mutation Positive Tumors Other Than MTC
Number analyzed (Participants) | 130 | 23 | 106 | 60 | 72 | 27 | 28 | 21 | 13
percentage of participants | 74.6 [66.2 to 81.8] | 78.3 [56.3 to 92.5] | 80.2 [71.3 to 87.3] | 80.0 [67.7 to 89.2] | 90.3 [81.0 to 96.0] | 85.2 [66.3 to 95.8] | 60.7 [40.6 to 78.5] | 28.6 [11.3 to 52.2] | 23.1 [5.0 to 53.8]

19. Secondary Outcome: Phase 2: DCR
Description: DCR was defined as the percentage of participants with a confirmed CR/PR, or SD, per RECIST v1.1. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in the short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in SOD of target lesions, taking as reference the smallest SOD on study (including baseline). DCR and its two-sided 95% CI, which is based on the exact binomial distribution (Clopper-Pearson), were presented.
Time Frame: Up to approximately 79.8 months
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment | RET-mutation MTC With Prior Cabozantinib and/or Vandetanib Treatment | RET-mutation MTC With No Prior Cabozantinib or Vandetanib Treatment | RET-fusion Positive TC | RET-fusion Positive Solid Tumors Other Than NSCLC and TC | RET-altered Solid Tumors Previously Treated With RET Inhibitor | RET-mutation Positive Tumors Other Than MTC
Number analyzed (Participants) | 130 | 23 | 106 | 60 | 72 | 27 | 28 | 21 | 13
percentage of participants | 91.5 [85.4 to 95.7] | 91.3 [72.0 to 98.9] | 89.6 [82.2 to 94.7] | 95.0 [86.1 to 99.0] | 93.1 [84.5 to 97.7] | 96.3 [81.0 to 99.9] | 75.0 [55.1 to 89.3] | 42.9 [21.8 to 66.0] | 69.2 [38.6 to 90.9]

20. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first dose of pralsetinib to the date of first documented PD or death due to any cause, whichever occurred first. PD was defined as at least a 20% increase in SOD of target lesions, taking as reference the smallest SOD on study (including baseline). PFS was analyzed using KM methods.
Time Frame: Up to approximately 7 years
Population: Efficacy population included all participants who have been exposed to at least one dose of the study drug at the RP2D. As pre-specified in the SAP, PFS was to be assessed in participants with RET-fusion positive NSCLC, RET-mutation MTC, RET-fusion TC, and RET-fusion solid tumors other than NSCLC and TC. Hence, only the data for these arms is presented here. Overall number analyzed is the number of participants with data available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment | RET-mutation MTC With Prior Cabozantinib and/or Vandetanib Treatment | RET-mutation MTC With No Prior Cabozantinib or Vandetanib Treatment | RET-fusion Positive TC | RET-fusion Positive Solid Tumors Other Than NSCLC and TC
Number analyzed (Participants) | 141 | 24 | 116 | 67 | 78 | 31 | 28
months | 16.4 [11.4 to 23.5] | 13.0 [9.3 to 35.1] | 12.1 [9.2 to 16.6] | 24.9 [19.9 to 35.0] | 55.3 [37.2 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [14.7 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 7.0 [3.9 to 12.8]

21. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time from the first dose of pralsetinib to the date of death due to any causes.
Time Frame: Up to approximately 7 years
Population: Efficacy population included all participants who have been exposed to at least one dose of the study drug at the RP2D. As pre-specified in the SAP, OS was to be assessed in participants with RET-fusion positive NSCLC, RET-mutation MTC, RET-fusion TC, and RET-fusion solid tumors other than NSCLC and TC. Hence, only the data for these arms is presented here.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment | RET-mutation MTC With Prior Cabozantinib and/or Vandetanib Treatment | RET-mutation MTC With No Prior Cabozantinib or Vandetanib Treatment | RET-fusion Positive TC | RET-fusion Positive Solid Tumors Other Than NSCLC and TC
Number analyzed (Participants) | 141 | 24 | 116 | 67 | 78 | 31 | 29
months | 39.7 [27.8 to 53.2] | 46.0 [19.1 to 62.4] | 50.1 [28.3 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 42.2 [31.2 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — The median and 95% CI was not estimable due to insufficient number of participants with events. | NA [19.4 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 10.3 [6.8 to 25.2]

22. Secondary Outcome: Phase 2: Intracranial ORR in RET-fusion Positive NSCLC Central Nervous System (CNS) Metastases Participants
Description: ORR=percentage of participants with CR or PR for at least 2 assessments with at least 28 days apart & no PD in between. CR=disappearance of all target CNS/brain lesion, including lesions in brain stem &/or cerebellum identified at baseline & disappearance of all non-target CNS/brain lesion at baseline & no identification of new CNS/brain lesion. PR =at least a 30% decrease in the SOD of any CNS/brain lesion, identified as RECIST 1.1 target lesions at baseline & if in the absence of unequivocal progression of any non-target CNS/brain lesion at baseline, or the identification of new CNS/brain lesion. PD=either at least 20% increase in the SOD of target CNS/brain lesion, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm or unequivocal progression of any CNS/brain lesion identified as RECIST 1.1 nontarget lesions at baseline, or the identification of new CNS/brain lesion.
Time Frame: Up to approximately 79.8 months
Population: RET-altered measurable disease population included participants in the efficacy population who have measurable (target) disease per RECIST v1.1, at baseline according to BICR and sufficient evidence of a RET alteration. As specified in the SAP, ORR was to be assessed in RET-fusion CNS metastases sub-population (participants with CNS metastases) only. Hence only NSCLC arms are presented here. Phase 1 participants treated at 400 mg QD are pooled with Phase 2 participants for efficacy analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment
Number analyzed (Participants) | 13 | 1 | 1
percentage of participants | 53.8 [25.1 to 80.8] | 100 [2.5 to 100] | 0 [NA to NA] — The 95% CI was not estimable due to insufficient number of participants with events.

23. Secondary Outcome: Phase 2: Intracranial CBR in RET-fusion Positive NSCLC CNS Metastases Participants
Description: CBR=percentage of participants with CR/PR/SD which has been lasting at least 16 weeks (i.e. 4 cycles if 28 days are in 1 cycle) from first dose date. CR=disappearance of all target CNS/brain lesion, including lesions in brain stem &/ cerebellum identified at baseline&disappearance of all non-target CNS/brain lesion at baseline & no identification of new CNS/brain lesion. PR=at least a 30% decrease in SOD of any CNS/brain lesion, identified as target lesions at baseline & if in absence of unequivocal progression of any non-target CNS/brain lesion at baseline, or identification of new CNS/brain lesion. SD=neither sufficient shrinkage for PR nor sufficient increase for PD for target/non-target CNS/brain lesion, taking as reference smallest SOD while on study. PD=either at least 20% increase in SOD of target CNS/brain lesion, taking as reference smallest sum on study. Unequivocal progression of any CNS/brain lesion nontarget lesions at baseline, or identification of new CNS/brain lesion.
Time Frame: Up to approximately 79.8 months
Population: RET-altered measurable disease population included participants in the efficacy population who have measurable (target) disease per RECIST v1.1, at baseline according to BICR and sufficient evidence of a RET alteration. As specified in the SAP, CBR was to be assessed in RET-fusion CNS metastases sub-population (participants with CNS metastases) only. Hence only NSCLC arms are presented here. Phase 1 participants treated at 400 mg QD are pooled with Phase 2 participants for efficacy analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment
Number analyzed (Participants) | 13 | 1 | 1
percentage of participants | 61.5 [31.6 to 86.1] | 100 [2.5 to 100] | 0 [NA to NA] — The 95% CI was not estimable due to insufficient number of participants with events.

24. Secondary Outcome: Phase 2: Intracranial DCR in RET-fusion Positive NSCLC CNS Metastases Participants
Description: DCR=percentage of participants with a confirmed CR/PR, or SD. CR=disappearance of all target CNS/brain lesion, including lesions in brain stem &/or cerebellum identified at baseline & disappearance of all non-target CNS/brain lesion at baseline & no identification of new CNS/brain lesion. PR =at least a 30% decrease in the SOD of any CNS/brain lesion, identified as RECIST 1.1 target lesions at baseline & if in the absence of unequivocal progression of any non-target CNS/brain lesion at baseline, or the identification of new CNS/brain lesion. SD=neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target/non-target CNS/brain lesion, taking as reference the smallest SOD while on study. PD=either at least 20% increase in SOD of target CNS/brain lesion, taking as reference smallest sum on study. Unequivocal progression of any CNS/brain lesion nontarget lesions at baseline, or identification of new CNS/brain lesion.
Time Frame: Up to approximately 79.8 months
Population: RET-altered measurable disease population included participants in the efficacy population who have measurable (target) disease per RECIST v1.1, at baseline according to BICR and sufficient evidence of a RET alteration. As specified in the SAP, DCR was to be assessed in RET-fusion CNS metastases sub-population (participants with CNS metastases) only. Hence only NSCLC arms are presented here. Phase 1 participants treated at 400 mg QD are pooled with Phase 2 participants for efficacy analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment
Number analyzed (Participants) | 13 | 1 | 1
percentage of participants | 76.9 [46.2 to 95.0] | 100 [2.5 to 100] | 0 [NA to NA] — The 95% CI was not estimable due to insufficient number of participants with events.

25. Secondary Outcome: Phase 2: Intracranial DOR in RET-fusion Positive NSCLC CNS Metastases Participants
Description: DOR=time from first documented CR/PR to the date of first documented PD/death due to any cause, whichever occurs first. CR=disappearance of all target CNS/brain lesion, including lesions in brain stem &/ cerebellum identified at baseline & disappearance of all non-target CNS/brain lesion at baseline & no identification of new CNS/brain lesion. PR=at least a 30% decrease in SOD of any CNS/brain lesion, identified as RECIST 1.1 target lesions at baseline & if in absence of unequivocal progression of any non-target CNS/brain lesion at baseline, or identification of new CNS/brain lesion. PD=either at least 20% increase in SOD of target CNS/brain lesion, taking as reference smallest sum on study. Unequivocal progression of any CNS/brain lesion nontarget lesions at baseline, or identification of new CNS/brain lesion. DOR was analyzed using the KM methods.
Time Frame: Up to approximately 79.8 months
Population: RET-altered measurable disease population=participants in efficacy population who have measurable (target) disease per RECIST v1.1, at baseline according to BICR&sufficient evidence of a RET alteration. As specified in SAP, DOR was to be assessed in RET-fusion CNS metastases sub-population only. Hence only NSCLC arms are presented here. Participants with a CR/PR were assessed for this OM. Phase 1 participants treated at 400 mg QD are pooled with Phase 2 participants for efficacy analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RET- Fusion Positive NSCLC With Prior Platinum Treatment | RET-fusion Positive NSCLC With Non-platinum Systemic Treatment | RET-fusion Positive NSCLC With No Prior Systemic or Platinum Treatment
Number analyzed (Participants) | 7 | 1 | 0
months | 28.3 [10.5 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 11.3 [NA to NA] — The 95% CI was not estimable due to insufficient number of participants with events. |

26. Secondary Outcome: Phase 1: Maximum Plasma Concentration (Cmax)
Description: Number of participants in each arm of this OM is based on the actual treatment received. 1 participant originally assigned to the 200/100 mg arm received the 100/100 mg treatment and hence, was counted under the 100/100 mg arm for this OM.
Time Frame: Predose on 0.5, 1, 2, 4, 6, 8 and 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: Pharmacokinetic (PK)-evaluable population included all participants who received at least one dose of pralsetinib and from whom at least one post dose PK sample was collected. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliters (ng/mL)
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg
Number analyzed (Participants) | 2 | 6 | 5 | 13 | 11 | 12 | 4 | 6 | 3
nanograms per milliliters (ng/mL)
  Cycle 1 Day 1 | 346 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 335 (52.8) | 198 (99.8) | 459 (52.3) | 688 (53.3) | 1210 (85.3) | 1820 (63.8) | 569 (42.0) | 715 (64.1)
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 6 | 3 | 12 | 9 | 10 | 2 | 5 | 2
  Cycle 1 Day 15 | 130 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. | 420 (56.9) | 586 (47.8) | 525 (72.5) | 1390 (35.3) | 1930 (66.7) | 4330 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 1080 (43.8) | 1780 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable.

27. Secondary Outcome: Phase 1: Time to Maximum Plasma Concentration (Tmax)
Description: as for outcome 26
Time Frame: Predose on 0.5, 1, 2, 4, 6, 8 and 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: PK evaluable population included all participants who received at least one dose of pralsetinib and from whom at least one post dose PK sample was collected. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Median (Full Range); unit: hour
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg
Number analyzed (Participants) | 2 | 6 | 5 | 13 | 11 | 12 | 4 | 6 | 3
hour
  Cycle 1 Day 1 | 3.04 [2.08 to 4.00] | 2.04 [1.98 to 4.00] | 2.03 [2.00 to 6.03] | 2.07 [0.983 to 7.98] | 2.02 [1.72 to 7.90] | 3.00 [2.00 to 6.03] | 2.00 [2.00 to 2.00] | 12.5 [12.2 to 14.8] | 12.0 [2.07 to 12.3]
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 6 | 3 | 12 | 9 | 10 | 2 | 5 | 2
  Cycle 1 Day 15 | 1.87 [1.87 to 1.87] | 2.00 [1.97 to 4.13] | 3.97 [3.90 to 4.00] | 2.97 [1.05 to 4.08] | 2.23 [0.983 to 24.0] | 3.03 [2.00 to 7.85] | 6.00 [4.00 to 8.00] | 2.00 [0.500 to 3.95] | 4.03 [1.98 to 6.08]

28. Secondary Outcome: Phase 1: Time of Last Quantifiable Plasma Drug Concentration (Tlast)
Description: The maximum values for Tlast slightly exceed 24 hours because the analysis used the actual time, i.e., the duration between dosing and actual sample collection, rather than the nominal sampling time of 24 hours specified in the protocol. The timeframe has been given as per nominal sampling timepoints pre-specified in the protocol. Number of participants in each arm of this OM is based on the actual treatment received. 1 participant originally assigned to the 200/100 mg arm received the 100/100 mg treatment and hence, was counted under the 100/100 mg arm for this OM.
Time Frame: Predose on 0.5, 1, 2, 4, 6, 8 and 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: as for outcome 27
Measure: Median (Full Range); unit: hours
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg
Number analyzed (Participants) | 2 | 6 | 5 | 13 | 11 | 12 | 4 | 6 | 3
hours
  Cycle 1 Day 1 | 24.0 [24.0 to 24.0] | 24.0 [23.1 to 24.4] | 24.0 [7.88 to 24.1] | 24.0 [21.9 to 25.7] | 23.8 [7.88 to 24.0] | 23.8 [22.6 to 24.6] | 23.9 [23.4 to 24.0] | 12.5 [12.2 to 14.8] | 12.3 [12.0 to 14.4]
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 6 | 3 | 12 | 9 | 10 | 2 | 5 | 2
  Cycle 1 Day 15 | 23.8 [23.8 to 23.8] | 24.1 [23.9 to 24.4] | 24.3 [23.6 to 27.8] | 24.0 [8.00 to 26.6] | 24.0 [22.2 to 24.8] | 24.0 [7.38 to 25.4] | 24.1 [24.0 to 24.2] | 12.2 [7.88 to 15.7] | 12.5 [10.1 to 14.8]

29. Secondary Outcome: Phase 1: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 24 Hours Postdose (AUC0-24)
Description: as for outcome 26
Time Frame: 24 hours postdose on Day 1 of Cycle 1 (1 cycle = 28 days)
Population: PK evaluable population included all participants who received at least one dose of pralsetinib and from whom at least one post dose PK sample was collected. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter (hours*ng/ml)
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg
Number analyzed (Participants) | 2 | 6 | 3 | 11 | 6 | 8 | 3 | 0 | 0
hours*nanograms/milliliter (hours*ng/ml) | 4450 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 3620 (50.8) | 3010 (84.8) | 5260 (46.2) | 8470 (54.5) | 14700 (60.3) | 27700 (94.1) |  |

30. Secondary Outcome: Phase 1: Plasma Drug Concentration at 24 Hours Postdose (C24hr)
Description: as for outcome 26
Time Frame: 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: PK evaluable population included all participants who received at least one dose of pralsetinib and from whom at least one post dose PK sample was collected. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg
Number analyzed (Participants) | 2 | 6 | 3 | 11 | 9 | 8 | 3 | 0 | 0
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 6 | 3 | 11 | 6 | 8 | 3 | 0 | 0
  Cycle 1 Day 1 | 110 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 69.2 (81.0) | 65.8 (59.6) | 104 (76.6) | 221 (64.2) | 376 (74.1) | 715 (75.9) |  |
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 6 | 3 | 10 | 9 | 8 | 2 | 0 | 0
  Cycle 1 Day 15 | 55.9 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. | 94.2 (123) | 175 (31.3) | 137 (132) | 713 (42.2) | 977 (107) | 1950 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. |  |

31. Secondary Outcome: Phase 1: Apparent Volume of Distribution (Vz/F)
Description: as for outcome 26
Time Frame: Predose on 0.5, 1, 2, 4, 6, 8 and 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg
Number analyzed (Participants) | 2 | 5 | 3 | 10 | 5 | 7 | 3 | 0 | 0
liters
  Cycle 1 Day 1 | 96.1 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 230 (37.1) | 458 (125) | 499 (50.8) | 543 (82.6) | 430 (62.6) | 350 (115) |  |
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 4 | 3 | 9 | 5 | 5 | 1 | 0 | 0
  Cycle 1 Day 15 | 355 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. | 171 (176) | 232 (43.7) | 622 (67.3) | 367 (86.6) | 418 (19.9) | 181 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. |  |

32. Secondary Outcome: Phase 1: Terminal Elimination Half-Life (t½)
Description: The maximum values for t1/2 slightly exceed 24 hours because the analysis used the actual time, i.e., the duration between dosing and actual sample collection, rather than the nominal sampling time of 24 hours specified in the protocol. The timeframe has been given as per nominal sampling timepoints pre-specified in the protocol. Number of participants in each arm of this OM is based on the actual treatment received. 1 participant originally assigned to the 200/100 mg arm received the 100/100 mg treatment and hence, was counted under the 100/100 mg arm for this OM.
Time Frame: Predose on 0.5, 1, 2, 4, 6, 8 and 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: as for outcome 30
Measure: Median (Full Range); unit: hours
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg
Number analyzed (Participants) | 2 | 5 | 3 | 10 | 5 | 7 | 3 | 0 | 1
hours
  Cycle 1 Day 1 | 16.3 [11.8 to 20.8] | 9.87 [8.98 to 18.3] | 14.3 [8.12 to 31.5] | 12.6 [6.69 to 34.9] | 12.2 [9.53 to 34.5] | 16.5 [10.2 to 48.7] | 19.7 [12.8 to 36.1] |  | 10.7 [10.7 to 10.7]
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 4 | 3 | 9 | 5 | 5 | 1 | 0 | 0
  Cycle 1 Day 15 | 17.6 [17.6 to 17.6] | 8.10 [5.25 to 39.6] | 13.4 [12.5 to 14.4] | 13.2 [10.1 to 21.8] | 20.4 [9.91 to 27.3] | 20.9 [9.21 to 33.6] | 13.0 [13.0 to 13.0] |  |

33. Secondary Outcome: Phase 1: Apparent Oral Clearance (CL/F)
Description: as for outcome 26
Time Frame: Predose on 0.5, 1, 2, 4, 6, 8 and 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/hr)
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg
Number analyzed (Participants) | 2 | 6 | 3 | 10 | 9 | 8 | 3 | 0 | 0
liters per hour (L/hr)
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 5 | 3 | 10 | 5 | 7 | 3 | 0 | 0
  Cycle 1 Day 1 | 4.26 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 14.7 (42.3) | 20.6 (48.1) | 27.3 (60.3) | 23.3 (40.2) | 15.2 (88.1) | 11.6 (81.3) |  |
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 6 | 3 | 10 | 9 | 8 | 2 | 0 | 0
  Cycle 1 Day 15 | 14.0 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. | 11.3 (51.2) | 12.0 (38.9) | 31.4 (97.8) | 13.2 (33.0) | 11.1 (72.2) | 8.57 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. |  |

34. Secondary Outcome: Phase 1: Accumulation Ratio for Cmax (RCmax)
Description: as for outcome 26
Time Frame: 24 hours postdose on Day 15 of Cycle 1 (1 cycle = 28 days)
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg
Number analyzed (Participants) | 1 | 6 | 3 | 12 | 9 | 10 | 2 | 4 | 1
ratio | 1.04 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. | 1.25 (27.6) | 3.20 (114) | 1.17 (110) | 1.87 (40.5) | 1.62 (102) | 2.97 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 1.91 (40.7) | 1.41 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable.

35. Secondary Outcome: Phase 1: Accumulation Ratio for AUC (RAUC)
Description: as for outcome 26
Time Frame: 24 hours postdose on Day 15 of Cycle 1 (1 cycle = 28 days)
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg
Number analyzed (Participants) | 1 | 6 | 1 | 8 | 4 | 6 | 1 | 2 | 1
ratio | 1.43 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. | 1.47 (11.1) | 3.22 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. | 1.31 (147) | 2.33 (11.4) | 2.75 (70.9) | 2.48 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. | 4.28 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 1.21 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable.

36. Secondary Outcome: Phase 2: Cmax
Time Frame: Predose on 0.5, 1, 2, 4, 6, 8 and 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- RET- Fusion Positive NSCLC Participants: Participants who had RET-fusion positive NSCLC received pralsetinib, 400 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons. This arm was specifically planned for reporting PK data.
- Tumor-agnostic Participants: Participants who had RET-fusion positive NSCLC or TC, or RET-mutation positive MTC, each with different genetic mutations received pralsetinib, 400 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons. This arm was specifically planned for reporting PK data.
- RET-altered Solid Tumors Participants: Participants who had RET-altered (fusion or mutation) solid tumors previously treated with a selective RET TKI received pralsetinib, 400 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons. This arm was specifically planned for reporting PK data.
- RET-mutation Positive Tumors Other Than MTC Participants: Participants who had RET-mutation positive solid tumors received Pralsetinib 400 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons. This arm was specifically planned for reporting PK data.
Arm/Group | RET- Fusion Positive NSCLC Participants | Tumor-agnostic Participants | RET-altered Solid Tumors Participants | RET-mutation Positive Tumors Other Than MTC Participants
Number analyzed (Participants) | 98 | 5 | 3 | 4
ng/mL
  Cycle 1 Day 1 | 1680 (69.4) | 1380 (65.4) | 2450 (164) | 1770 (87.2)
  Cycle 1 Day 15: number analyzed (Participants) | 87 | 5 | 3 | 4
  Cycle 1 Day 15 | 2840 (50.7) | 2200 (36.7) | 3440 (93.9) | 2430 (55.3)

37. Secondary Outcome: Phase 2: Tmax
Time Frame: Predose on 0.5, 1, 2, 4, 6, 8 and 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: as for outcome 30
Measure: Median (Full Range); unit: hours
Arm/Group | RET- Fusion Positive NSCLC Participants | Tumor-agnostic Participants | RET-altered Solid Tumors Participants | RET-mutation Positive Tumors Other Than MTC Participants
Number analyzed (Participants) | 98 | 5 | 3 | 4
hours
  Cycle 1 Day 1 | 4.00 [1.90 to 23.7] | 3.90 [2.0 to 6.0] | 4.0 [4.0 to 6.0] | 2.05 [2 to 8]
  Cycle 1 Day 15: number analyzed (Participants) | 87 | 5 | 3 | 4
  Cycle 1 Day 15 | 4.00 [1.00 to 8.10] | 5.00 [2.0 to 8.0] | 4.00 [2.00 to 6.00] | 3.05 [2 to 6]

38. Secondary Outcome: Phase 2: Tlast
Description: The maximum values for Tlast slightly exceed 24 hours because the analysis used the actual time, i.e., the duration between dosing and actual sample collection, rather than the nominal sampling time of 24 hours specified in the protocol. The timeframe has been given as per nominal sampling timepoints pre-specified in the protocol.
Time Frame: Predose on 0.5, 1, 2, 4, 6, 8 and 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: as for outcome 30
Measure: Median (Full Range); unit: hours
Arm/Group | RET- Fusion Positive NSCLC Participants | Tumor-agnostic Participants | RET-altered Solid Tumors Participants | RET-mutation Positive Tumors Other Than MTC Participants
Number analyzed (Participants) | 98 | 5 | 3 | 4
hours
  Cycle 1 Day 1 | 23.9 [2.40 to 24.8] | 8.00 [7.8 to 23.5] | 23.10 [8.0 to 24.0] | 8.05 [8.0 to 24.0]
  Cycle 1 Day 15: number analyzed (Participants) | 87 | 5 | 3 | 4
  Cycle 1 Day 15 | 23.8 [7.80 to 26.5] | 23.70 [7.9 to 24.0] | 24.00 [7.9 to 24.0] | 24.00 [23.8 to 24.0]

39. Secondary Outcome: Phase 2: AUC0-24
Time Frame: 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | RET- Fusion Positive NSCLC Participants | Tumor-agnostic Participants | RET-altered Solid Tumors Participants | RET-mutation Positive Tumors Other Than MTC Participants
Number analyzed (Participants) | 70 | 3 | 2 | 4
hours*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 70 | 2 | 1 | 3
  Cycle 1 Day 1 | 20400 (64.2) | 17400 (152) | 103000 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. | 18400 (69.8)
  Cycle 1 Day 15: number analyzed (Participants) | 50 | 3 | 2 | 4
  Cycle 1 Day 15 | 40100 (59.5) | 33900 (27.4) | 91100 (46.8) | 32000 (90.8)

40. Secondary Outcome: Phase 2: C24hr
Time Frame: 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | RET- Fusion Positive NSCLC Participants | Tumor-agnostic Participants | RET-altered Solid Tumors Participants | RET-mutation Positive Tumors Other Than MTC Participants
Number analyzed (Participants) | 92 | 5 | 3 | 4
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 92 | 5 | 3 | 3
  Cycle 1 Day 1 | 540 (75.4) | 519 (197) | 1020 (225) | 415 (140)
  Cycle 1 Day 15: number analyzed (Participants) | 82 | 5 | 2 | 4
  Cycle 1 Day 15 | 1150 (69) | 797 (42.8) | 1400 (207) | 1050 (94.0)

41. Secondary Outcome: Phase 2: t½
Description: The maximum values for t1/2 slightly exceed 24 hours because the analysis used the actual time, i.e., the duration between dosing and actual sample collection, rather than the nominal sampling time of 24 hours specified in the protocol. The timeframe has been given as per nominal sampling timepoints pre-specified in the protocol.
Time Frame: Predose on 0.5, 1, 2, 4, 6, 8 and 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- RET- Fusion Positive NSCLC Participants: Participants who had RET-fusion positive NSCLC received pralsetinib, 400 mg orally, QD until discontinuation due to toxicity, disease progression, or other reasons. This arm was specifically planned for reporting PK data. This arm was specifically planned for reporting PK data.
- RET-mutation Positive Tumors Other Than MTC Participants: Participants who had RET-mutation positive solid tumors received Pralsetinib 400 mg, orally, QD until discontinuation due to toxicity, disease progression, or other reasons. This arm was specifically planned for reporting PK data. This arm was specifically planned for reporting PK data.
Arm/Group | RET- Fusion Positive NSCLC Participants | Tumor-agnostic Participants | RET-altered Solid Tumors Participants | RET-mutation Positive Tumors Other Than MTC Participants
Number analyzed (Participants) | 57 | 2 | 1 | 3
hours
  Cycle 1 Day 1 | 13.4 (44.1) | 18.4 (98.8) | 20.8 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. | 11.0 (55.8)
  Cycle 1 Day 15: number analyzed (Participants) | 47 | 2 | 1 | 2
  Cycle 1 Day 15 | 17.9 (58.8) | 16.5 (44.6) | 25.8 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. | 63.0 (882)

42. Secondary Outcome: Phase 2: CL/F
Time Frame: Predose on 0.5, 1, 2, 4, 6, 8 and 24 hours postdose on Days 1 and 15 of Cycle 1 (1 cycle = 28 days)
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/hour)
Arm/Group | RET- Fusion Positive NSCLC Participants | Tumor-agnostic Participants | RET-altered Solid Tumors Participants | RET-mutation Positive Tumors Other Than MTC Participants
Number analyzed (Participants) | 47 | 2 | 1 | 3
liters per hour (L/hour)
  Cycle 1 Day 1: number analyzed (Participants) | 30 | 2 | 1 | 3
  Cycle 1 Day 1 | 13.4 (56.8) | 12.7 (347) | 2.00 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. | 16.1 (43.3)
  Cycle 1 Day 15: number analyzed (Participants) | 47 | 2 | 1 | 2
  Cycle 1 Day 15 | 9.91 (58.9) | 7.49 (64.4) | 2.92 (NA) — Since data was available only for 1 participant geometric co-efficient of variation was not evaluable. | 1.39 (1220)

43. Secondary Outcome: Phase 1: Percent Change From Baseline in Dual Specificity Phosphatase 6 (DUSP6)
Description: The dose dependent change in a mitogen-activated protein kinases (MAPK) pathway expression signature was analyzed for all available samples of MTC and NSCLC participants. Participants with archived sample (used as baseline) and on treatment Cycle 2 Day 1 (1 cycle = 28 days) tumor tissues with greater than 20% tumor cells are included in the analysis. The changes in tumor biomarker DUSP6 levels was explored.
Time Frame: Baseline, Week 4
Population: Safety Population included all participants who have received at least 1 dose of the study drug regardless of starting dose levels.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg
Number analyzed (Participants) | 2 | 6 | 5 | 13 | 11 | 12 | 4 | 5 | 4
percent change | 0 (0) | 54.26 (88.318) | 0 (0) | -20.27 (42.971) | -74.87 (15.707) | -13.32 (82.394) | 0 (0) | -81.57 (3.057) | -61.96 (39.141)

44. Secondary Outcome: Phase 1: Percent Change From Baseline in Sprout Receptor Tyrosine Kinase Signaling Antagonist 4 (SPRY4)
Description: The dose dependent change in a MAPK pathway expression signature was analyzed for all available samples of MTC and NSCLC participants. Participants with archived sample (used as baseline) and on treatment Cycle 2 Day 1 (1 cycle = 28 days) tumor tissues with greater than 20% tumor cells are included in the analysis. The changes in tumor biomarker SPRY4 levels was explored.
Time Frame: Baseline, Week 4
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase I: Pralsetinib 30 mg | Phase I: Pralsetinib 60 mg | Phase I: Pralsetinib 100 mg | Phase I: Pralsetinib 200 mg | Phase I: Pralsetinib 300 mg | Phase I: Pralsetinib 400 mg | Phase I: Pralsetinib 600 mg | Phase I: Pralsetinib 100/100 mg | Phase I: Pralsetinib 200/100 mg
Number analyzed (Participants) | 2 | 6 | 5 | 13 | 11 | 12 | 4 | 5 | 4
percent change | 0 (0) | 210.16 (309.468) | 0 (0) | -34.98 (29.569) | -69.00 (28.731) | -3.26 (99.349) | 0 (0) | -75.65 (10.944) | 124.93 (311.210)

ADVERSE EVENTS:
Time Frame: AEs and SAEs: From Cycle 1 Day 1 up to 30 days after the final dose of study drug (up to approximately 6.7 years) All-cause Mortality: Up to approximately 7 years Safety population included all participants who have received at least 1 dose of the study drug regardless of starting dose levels.
Description: As pre-specified in SAP, safety data was to be analyzed & reported per pre-planned grouped dose level II. Per dose level II, ≤ 300 mg QD arm included participants dosed with pralsetinib at 30 mg, 60 mg , 100 mg , 200 mg & 300 mg QD; 400 mg arm included participants dosed at 400 mg QD, BID Dosing Schedule arm included participants dosed with 100/100 mg & 200/100 mg BID, & All doses included participants treated at all QD & BID doses & 600 mg QD dose. Hence, AEs cannot be presented per dose level.
Arm/Group | Pralsetinib ≤ 300 mg QD | Pralsetinib 400 mg QD | Pralsetinib BID Dosing Schedule | Pralsetinib All Doses
All-Cause Mortality (participants affected / at risk) | 15/37 | 245/540 | 7/9 | 268/590
Serious Adverse Events (participants affected / at risk) | 26/37 | 381/540 | 7/9 | 416/590
Other Adverse Events (participants affected / at risk) | 36/37 | 536/540 | 9/9 | 585/590
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pralsetinib ≤ 300 mg QD (N=37) | Pralsetinib 400 mg QD (N=540) | Pralsetinib BID Dosing Schedule (N=9) | Pralsetinib All Doses (N=590)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 32 (50) | 1 (1) | 34 (52)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Eosinophilia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (6) | 0 (0) | 5 (6)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 8 (11) | 0 (0) | 8 (11)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (62) | 0 (0) | 2 (62)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Myocardial injury (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (2) | 3 (3) | 0 (0) | 4 (5)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 7 (7) | 1 (1) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 6 (8) | 0 (0) | 6 (8)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (6) | 0 (0) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 7 (7) | 0 (0) | 9 (9)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 7 (7) | 1 (1) | 8 (8)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (4)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 3 (4)
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 3 (5) | 0 (0) | 3 (5)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Proctitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (6) | 0 (0) | 3 (6)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 5 (5) | 0 (0) | 7 (8)
Asthenia (General disorders) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Calcinosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 6 (6) | 0 (0) | 6 (6)
Disease progression (General disorders) | 0 (0) | 10 (10) | 0 (0) | 10 (10)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (4) | 0 (0) | 4 (5)
General physical health deterioration (General disorders) | 0 (0) | 4 (5) | 0 (0) | 4 (5)
Granuloma (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Performance status decreased (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 15 (21) | 0 (0) | 15 (21)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 7 (8) | 0 (0) | 8 (9)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (4)
Subcapsular hepatic haematoma (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Atypical mycobacterial pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 8 (8) | 0 (0) | 9 (9)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 16 (18) | 0 (0) | 17 (19)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 13 (18) | 0 (0) | 14 (19)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 4 (4)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (3) | 3 (3) | 0 (0) | 4 (6)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 6 (6)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatitis B reactivation (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Klebsiella urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymph node tuberculosis (Infections and infestations) | 0 (0) | 2 (4) | 0 (0) | 2 (4)
Meningitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Meningitis enterococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pancreatic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 5 (6) | 0 (0) | 6 (7)
Pneumonia (Infections and infestations) | 5 (5) | 87 (120) | 1 (1) | 94 (127)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 3 (5) | 0 (0) | 3 (5)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Scrotal cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 20 (23) | 3 (5) | 25 (30)
Septic arthritis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Sinusitis aspergillus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Spontaneous bacterial peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 3 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 23 (40) | 1 (1) | 26 (43)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (7) | 0 (0) | 4 (7)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 2 (7) | 0 (0) | 2 (7)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 0 (0) | 3 (4)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (4) | 0 (0) | 3 (4)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 5 (5) | 0 (0) | 5 (5)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Inflammatory marker increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 4 (15) | 0 (0) | 4 (15)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (4)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 0 (0) | 3 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (8) | 0 (0) | 5 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 8 (14) | 1 (1) | 10 (16)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 0 (0) | 3 (5)
Pseudohyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (8) | 0 (0) | 8 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (11) | 0 (0) | 9 (11)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (4)
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (3) | 2 (4)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 26 (30) | 0 (0) | 27 (31)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 0 (0) | 5 (5)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 6 (6) | 0 (0) | 6 (6)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 7 (7) | 0 (0) | 7 (7)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) | 3 (4)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 5 (6) | 0 (0) | 5 (6)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (4)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malignant spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Polyneuropathy chronic (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 7 (10) | 0 (0) | 7 (10)
Syncope (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Vertebral artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Device issue (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 3 (4) | 0 (0) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 5 (6) | 0 (0) | 6 (7)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Obstructive nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 1 (1) | 6 (6)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 10 (14) | 0 (0) | 10 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (12) | 0 (0) | 6 (12)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 11 (12) | 1 (1) | 14 (15)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 27 (32) | 0 (0) | 29 (35)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (7) | 0 (0) | 6 (8)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8) | 0 (0) | 12 (12)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7) | 1 (1) | 9 (10)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 8 (9) | 0 (0) | 8 (9)
Hypotension (Vascular disorders) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Internal haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pralsetinib ≤ 300 mg QD (N=37) | Pralsetinib 400 mg QD (N=540) | Pralsetinib BID Dosing Schedule (N=9) | Pralsetinib All Doses (N=590)
Anaemia (Blood and lymphatic system disorders) | 16 (45) | 285 (1098) | 6 (15) | 310 (1168)
Leukopenia (Blood and lymphatic system disorders) | 4 (11) | 55 (226) | 1 (1) | 61 (239)
Lymphopenia (Blood and lymphatic system disorders) | 7 (29) | 67 (321) | 2 (8) | 77 (359)
Neutropenia (Blood and lymphatic system disorders) | 8 (22) | 124 (422) | 2 (6) | 135 (456)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (6) | 44 (98) | 1 (1) | 48 (105)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Corneal epithelial microcysts (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye disorder (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Growth of eyelashes (Eye disorders) | 0 (0) | 4 (4) | 1 (1) | 5 (5)
Vision blurred (Eye disorders) | 1 (1) | 34 (49) | 1 (1) | 37 (52)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 9 (11) | 0 (0) | 11 (13)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 27 (33) | 0 (0) | 29 (35)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 68 (89) | 0 (0) | 74 (95)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 46 (56) | 2 (2) | 49 (59)
Ascites (Gastrointestinal disorders) | 1 (1) | 19 (31) | 2 (2) | 23 (35)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 5 (5)
Constipation (Gastrointestinal disorders) | 12 (16) | 238 (329) | 2 (2) | 255 (351)
Diarrhoea (Gastrointestinal disorders) | 10 (19) | 189 (373) | 4 (7) | 207 (407)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 92 (103) | 1 (1) | 96 (110)
Dyspepsia (Gastrointestinal disorders) | 3 (5) | 29 (36) | 0 (0) | 32 (41)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 44 (50) | 1 (1) | 47 (53)
Gastritis (Gastrointestinal disorders) | 0 (0) | 10 (10) | 1 (1) | 11 (11)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 34 (41) | 2 (2) | 37 (44)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 13 (17) | 2 (2) | 15 (19)
Nausea (Gastrointestinal disorders) | 10 (17) | 114 (163) | 1 (1) | 126 (182)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 33 (53) | 0 (0) | 37 (57)
Toothache (Gastrointestinal disorders) | 0 (0) | 14 (15) | 1 (1) | 15 (16)
Vomiting (Gastrointestinal disorders) | 7 (10) | 88 (113) | 0 (0) | 95 (123)
Asthenia (General disorders) | 1 (1) | 88 (192) | 0 (0) | 90 (194)
Calcinosis (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Chest discomfort (General disorders) | 1 (1) | 16 (19) | 1 (1) | 18 (21)
Chills (General disorders) | 4 (4) | 28 (30) | 0 (0) | 32 (34)
Face oedema (General disorders) | 1 (1) | 42 (57) | 0 (0) | 43 (58)
Fatigue (General disorders) | 12 (17) | 154 (289) | 2 (2) | 169 (309)
Localised oedema (General disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Malaise (General disorders) | 0 (0) | 33 (44) | 0 (0) | 34 (45)
Mucosal inflammation (General disorders) | 3 (4) | 40 (56) | 0 (0) | 43 (60)
Non-cardiac chest pain (General disorders) | 4 (4) | 21 (22) | 2 (2) | 27 (28)
Oedema peripheral (General disorders) | 9 (10) | 104 (140) | 4 (4) | 117 (154)
Peripheral swelling (General disorders) | 4 (5) | 17 (19) | 1 (1) | 22 (25)
Pyrexia (General disorders) | 7 (11) | 164 (266) | 3 (7) | 176 (286)
Bronchitis (Infections and infestations) | 1 (2) | 23 (28) | 1 (1) | 25 (31)
COVID-19 (Infections and infestations) | 2 (4) | 64 (71) | 0 (0) | 66 (75)
Cellulitis (Infections and infestations) | 1 (1) | 9 (10) | 1 (1) | 12 (13)
Ear infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Folliculitis (Infections and infestations) | 0 (0) | 6 (6) | 1 (2) | 7 (8)
Fungal foot infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 13 (14) | 1 (1) | 15 (16)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 7 (7)
Oral candidiasis (Infections and infestations) | 2 (2) | 17 (26) | 1 (1) | 21 (30)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Pneumonia (Infections and infestations) | 4 (4) | 64 (107) | 0 (0) | 68 (111)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 3 (5) | 18 (18) | 1 (1) | 22 (24)
Skin candida (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 51 (61) | 1 (1) | 53 (63)
Urinary tract infection (Infections and infestations) | 5 (10) | 80 (167) | 1 (4) | 87 (182)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 18 (21) | 2 (3) | 21 (26)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Alanine aminotransferase increased (Investigations) | 16 (31) | 212 (459) | 3 (4) | 232 (495)
Aspartate aminotransferase increased (Investigations) | 17 (41) | 273 (693) | 3 (3) | 295 (739)
Blood alkaline phosphatase increased (Investigations) | 8 (9) | 68 (112) | 1 (1) | 78 (125)
Blood bilirubin increased (Investigations) | 2 (5) | 58 (166) | 1 (1) | 61 (172)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 97 (445) | 0 (0) | 97 (445)
Blood creatinine increased (Investigations) | 11 (17) | 143 (288) | 3 (4) | 158 (310)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 47 (72) | 0 (0) | 47 (72)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 31 (39) | 0 (0) | 32 (40)
Electrocardiogram repolarisation abnormality (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 38 (108) | 0 (0) | 38 (108)
Hepatic enzyme increased (Investigations) | 2 (4) | 2 (4) | 1 (1) | 5 (9)
Lymphocyte count decreased (Investigations) | 6 (18) | 90 (345) | 1 (3) | 98 (379)
Neutrophil count decreased (Investigations) | 5 (16) | 146 (539) | 1 (1) | 153 (558)
Platelet count decreased (Investigations) | 3 (5) | 67 (166) | 0 (0) | 72 (173)
Weight decreased (Investigations) | 2 (2) | 36 (50) | 0 (0) | 38 (52)
Weight increased (Investigations) | 2 (4) | 62 (170) | 0 (0) | 64 (174)
White blood cell count decreased (Investigations) | 14 (41) | 157 (579) | 2 (3) | 175 (636)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 113 (164) | 3 (3) | 124 (175)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 10 (12) | 0 (0) | 12 (14)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (3) | 21 (32) | 1 (1) | 24 (36)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 37 (59) | 0 (0) | 39 (61)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 29 (50) | 1 (1) | 33 (54)
Hyperphosphataemia (Metabolism and nutrition disorders) | 4 (4) | 101 (177) | 3 (4) | 109 (186)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (6) | 84 (228) | 0 (0) | 89 (234)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (12) | 130 (321) | 1 (3) | 138 (336)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (19) | 98 (163) | 1 (3) | 103 (185)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (5) | 54 (105) | 0 (0) | 58 (110)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 70 (122) | 3 (6) | 79 (135)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (16) | 75 (131) | 3 (4) | 84 (151)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 90 (118) | 3 (3) | 100 (130)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 88 (119) | 1 (1) | 95 (126)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 42 (50) | 0 (0) | 46 (54)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 19 (23) | 0 (0) | 21 (25)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 67 (121) | 0 (0) | 69 (123)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 34 (39) | 0 (0) | 36 (41)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 66 (105) | 0 (0) | 72 (111)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (8) | 1 (1) | 6 (9)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (6) | 1 (2) | 5 (8)
Dizziness (Nervous system disorders) | 7 (9) | 83 (101) | 2 (2) | 94 (115)
Dysgeusia (Nervous system disorders) | 2 (4) | 74 (97) | 0 (0) | 77 (102)
Headache (Nervous system disorders) | 8 (8) | 100 (140) | 1 (1) | 110 (152)
Hypoaesthesia (Nervous system disorders) | 5 (5) | 35 (46) | 0 (0) | 40 (51)
Memory impairment (Nervous system disorders) | 1 (1) | 13 (18) | 1 (1) | 15 (20)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 26 (36) | 0 (0) | 32 (43)
Paraesthesia (Nervous system disorders) | 0 (0) | 33 (35) | 0 (0) | 33 (35)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 21 (26) | 1 (1) | 22 (27)
Anxiety (Psychiatric disorders) | 4 (4) | 28 (31) | 0 (0) | 32 (35)
Depression (Psychiatric disorders) | 2 (2) | 19 (20) | 0 (0) | 21 (22)
Insomnia (Psychiatric disorders) | 2 (2) | 47 (56) | 2 (2) | 52 (61)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 17 (21) | 1 (1) | 19 (23)
Dysuria (Renal and urinary disorders) | 1 (1) | 28 (34) | 0 (0) | 29 (35)
Renal failure (Renal and urinary disorders) | 1 (1) | 8 (9) | 1 (2) | 10 (12)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Breast calcifications (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2) | 30 (34) | 0 (0) | 32 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 149 (222) | 2 (2) | 161 (236)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 47 (55) | 1 (1) | 49 (57)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 112 (146) | 2 (3) | 127 (165)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 22 (32) | 1 (1) | 24 (34)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 41 (49) | 0 (0) | 43 (51)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 19 (22) | 1 (1) | 24 (27)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 41 (54) | 0 (0) | 45 (58)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 16 (36) | 0 (0) | 18 (38)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 51 (97) | 1 (1) | 59 (109)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 35 (39) | 1 (1) | 36 (40)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 1 (1) | 7 (7)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 1 (1) | 4 (5)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 34 (37) | 0 (0) | 37 (40)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 17 (18) | 2 (2) | 22 (23)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 21 (25) | 1 (1) | 25 (29)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (10) | 0 (0) | 11 (12)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (4) | 16 (20) | 1 (1) | 19 (25)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 58 (71) | 0 (0) | 61 (74)
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 0 (0) | 8 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 14 (16) | 1 (1) | 15 (17)
Haematoma (Vascular disorders) | 0 (0) | 6 (6) | 1 (1) | 7 (7)
Hypertension (Vascular disorders) | 9 (12) | 189 (499) | 4 (11) | 206 (530)
Hypotension (Vascular disorders) | 2 (2) | 13 (16) | 0 (0) | 15 (18)
Intermittent claudication (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Vasodilatation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT03037385/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT03037385/SAP_001.pdf